CLINICAL TRIAL: NCT01139814
Title: Clinical Study to Evaluate the Effectiveness and Safety of the Catheter Robotics Amigo Remote Catheter System for Performing Right-Sided Electrophysiology Mapping Studies
Brief Title: Clinical Study to Evaluate the Catheter Robotics Amigo for Performing Right-Sided Electrophysiology Mapping Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catheter Robotics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-001-01
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Results first posted 2013-04-10 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Atrial Flutter; Ventricular Tachycardia
Keywords: atrial flutter; AVNRT; right sided accessory pathway; ventricular tachycardia; Patients who have one or more standard indications for a right-sided diagnostic electrophysiology procedure.
MeSH Terms: conditions — Atrial Flutter; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Catheter Robot (Experimental): device
  Interventions: Device: Amigo catheter robot

INTERVENTIONS:
Device: Amigo catheter robot — The Amigo Catheter System is intended to facilitate manipulation, positioning and control of a Diagnostic Catheter.

SUMMARY:
The purpose of this clinical study is to collect safety and performance data to support a demonstration of substantial equivalence of the Catheter Robotics Remote Catheter System to predicate devices when used to perform EP mapping of the right heart (atrium and ventricle).

ELIGIBILITY:
Inclusion Criteria:

1. > 18years of age.
2. Indicated for a right-sided electrophysiology ablation study (e.g., atrial flutter, AVNRT, right-sided accessory pathway, or ventricular tachycardia).
3. Willingness, ability, and commitment to participate in the procedure visit and a follow-up evaluation including a clinic visit at 7 (-0, +7) days after the study procedure.
4. Completion of Informed Consent.

Exclusion Criteria:

1. Any contraindication to cardiac catheterization, including pregnancy.
2. Enrollment in any other ongoing cardiac device trial.
3. Right-sided cardiac prosthetics including implanted active energy devices with permanent leads in or through the right atrium and/or ventricle.
4. Corrected or uncorrected atrial septal defect (ASD).
5. Poor general health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e., other disease processes, mental capacity, etc.).
6. Medical condition that will require anticoagulation during study or ablation procedure.
7. Presence of atrial fibrillation or atrial flutter at time of study procedure.
8. Other condition observed prior to the procedure where, in the view of the physician, participation in the study could further present a risk to the subject.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Sequoia Hospital, Redwood City, California
  - Northwestern Medical Center, Chicago, Illinois
  - Genesis Health,, Davenport, Iowa
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Gagnon Cardiovascular Institute/Morristown Memorial Hospital, Morristown, New Jersey
  - Lenox Hill Hospital, New York, New York
  - Lancaster Heart & Stroke Foundation, Lancaster, Pennsylvania
  - Lone Star Heart Center, Amarillo, Texas
  - Valley Health, Winchester, Virginia
- Glenfield Hospital, Leicester, United Kingdom

REFERENCES:
- [Derived] Khan EM, Frumkin W, Ng GA, Neelagaru S, Abi-Samra FM, Lee J, Giudici M, Gohn D, Winkle RA, Sussman J, Knight BP, Berman A, Calkins H. First experience with a novel robotic remote catheter system: Amigo mapping trial. J Interv Card Electrophysiol. 2013 Aug;37(2):121-9. doi: 10.1007/s10840-013-9791-9. Epub 2013 May 1. PMID 23636870

RESULTS

PARTICIPANT FLOW:
Groups:
- Intent-to-Treat: Subject was evaluated for the study criteria on the day of procedure, Investigator positioned the mapping catheter in the right heart, and connected the mapping catheter to the Amigo RCS.
  Amigo RCS is an accessory for use in the cardiac EP setting to allow the operator to manipulate a steerable cardiac catheter and perform a conventional electrophysiology procedure. The intent of the device is to allow the operator to complete the procedure in a conventional x-ray guided EP lab. Catheter control can be performed while standing (or sitting) some distance from the subject to minimize absorbed radiology dose and minimize operator fatigue from standing for long periods of time with the standard lead aprons/personal protection devices.
Period: Overall Study
Arm/Group | Intent-to-Treat
Started | 181
Completed | 181
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intent-to-Treat: Subject was evaluated for the study criteria on the day of procedure, Investigator positioned the mapping catheter in the right heart, and connected the mapping catheter to the Amigo RCS.
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 181
Age Continuous [Mean (Standard Deviation); unit: years] | 56.6 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 81
Region of Enrollment [Number; unit: participants]
  United States | 152
  United Kingdom | 29

OUTCOME MEASURES:

1. Primary Outcome: Navigation Performance
Description: Effectiveness Navigation Performance -- The ability to navigate the mapping catheter under Amigo control to at least 80% of 8 pre-specified anatomical locations over all subjects.
Time Frame: During Procedure
Measure: Number (95% Confidence Interval); unit: Successful locations
Units Other Than Participants: Locations
Groups:
- Intent-to-Treat: A subject was considered Intent-to-treat once the subject was evaluated for the study criteria on the day of procedure, the Investigator positioned the mapping catheter in the right heart, and connected the mapping catheter to the Amigo RCS.
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 181
Number analyzed (Locations) | 1448
Successful locations | 1396 [1370 to 1422]

2. Primary Outcome: Evaluation of Major Complications
Description: Safety Evaluation of Major Complications definitely or probably related to Amigo-Controlled Mapping through Visit 3 follow-up.
Time Frame: Seven Days (visit 3), except for any subject with an ongoing SAE that is related to the study will be scheduled for additional evaluations at 14 day intervals.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Intent-to-Treat
Number analyzed (Participants) | 181
Participants | 0 [0 to 4]

ADVERSE EVENTS:
Time Frame: Evaluation of adverse events definitely or probably related to Amigo RCS controlled mapping through 7 day follow-up.
Description: Only adverse events related to the device are posted
Arm/Group | Intent-to-Treat
Serious Adverse Events (participants affected / at risk) | 0/181
Other Adverse Events (participants affected / at risk) | 1/181
OTHER ADVERSE EVENTS (reported when occurring in more than 0.55% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-Treat (N=181)
Atrial Tachycardia (Cardiac disorders) | 1 (1) — Subject experienced SVT during mapping with Amigo. Attempts were made to terminate arrhythmia but a right bundle morphology was seen for the rest of the procedure. The CEC adjudicated the event as non serious, minor and probably related to device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less